CLINICAL TRIAL: NCT02619123
Title: Tailored Screening for Breast Cancer in Premenopausal Women. A Translational, Randomized Population-based Trial
Brief Title: Tailored Screening for Breast Cancer in Premenopausal Women
Acronym: TBST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Prevention and Research Institute, Italy (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: RF-2009-1493239
Record Dates: First submitted 2015-11-12; First posted 2015-12-02 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: breast density; breast cancer; risk-based screening; Tailored breast cancer screening; premenopausal women
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- invitation to mammography screening (Active Comparator): 44-45 years old women in this arm are invited to attend for a mammography screening every 1 year. After the age of 50, all women will continue to be screened in the usual service screening programme.
  Interventions: Other: Annual invitation to mammography
- invitation to tailored screening (Experimental): 44-45 years old women in this arm with a dense breast (3-4 categories in BI-RADS) at the baseline mammography are invited again after 1 year, while the lower-density group in the intervention arm are invited after 2 years. After the age of 50, all women will continue to be screened in the usual service screening programme.
  Interventions: Other: Tailored screening according to breast density

INTERVENTIONS:
Other: Tailored screening according to breast density — Different interval of mammography screening according to breast density
  Arms: invitation to tailored screening
Other: Annual invitation to mammography — Annual interval mammography screening according to international guidelines for women younger than 50 years old
  Arms: invitation to mammography screening

SUMMARY:
The Tailored Breast Screening Trial (TBST) is a population-based, non-inferiority randomised trial aimed at evaluating the impact of tailored screening strategies addressed to premenopausal women, by using breast density as indicator of risk.

44-45 years old women will be enrolled and invited to undergo a digital mammography. Women are then randomly allocated in two arms. In the intervention arm, women will receive a tailored screening strategy according to breast density.

The aim of this study is to assess the impact of a longer screening interval and the reduction of side effects for premenopausal women.

DETAILED DESCRIPTION:
Introduction: the Tailored Breast Screening Trial (TBST) is a population-based, non-inferiority randomised trial aimed at evaluating the impact of a change in the screening protocol in a service screening practice. "Tailored" means that the use of a breast density classification allocates women to a longer interval, decreasing the number of screening rounds in the 45-50-year age range. Density of the breast at the baseline is considered as an indicator of risk and also as a masking factor. The aim of this study is to assess the impact of a longer interval and the reduction of side effects for women allocated to the intervention group. In this study, any further intervention is offered to high-density women who are followed-up according to the usual care interval, since the study aimed at decreasing the screening burden.

Methods 44- 45 years old women resident in the screening centre catchment area will be invited to attend for mammography screening and will be asked for informed consent in order to be included in the study. After the enrolment, they will receive a high quality digital mammography; two views and breast density will be classified according with the BI-RADS classification. Women are randomly allocated either to an usual care group or to the intervention group. In the intervention group, women with a dense breast (3-4 categories in BI-RADS) will be invited again after 1 year, while the lower-density group in the intervention arm will be invited after 2 years. After the age of 50, all women will continue to be screened in the usual service screening programme. Density of the breast will be read by 2 readers, and controversies will be solved by a consensus. Allocation of women is blinded to the mammography readers.

EXPECTED RESULTS: the outcomes are: 1. cumulative incidence of interval-cancer cases by intention to treat grouping and by density group, aimed at assessing the non inferiority of screening performance; 2. cumulative incidence of T2+/node-positive status breast cancer cases between arms and by protocol. Screening performance parameters will be evaluated at each screening round. Interim and outcome analysis are expected at 3 and 6 years average follow-up, respectively, starting from the beginning of the screening.

SAMPLE SIZE: the non-inferiority limit is derived from the accepted level of interval cancers in women 50-69 years, which was considered acceptable by the European Community Guidelines. Assuming a 70%BI-RADS 1-2 at the baseline on the basis of the digital mammography experience, the estimated sample size with a power of 90% is 16,596 women per arm.

ELIGIBILITY:
Inclusion Criteria:

* women 44-45 years old resident in the screening area

Exclusion Criteria:

* previous diagnosis of invasive or in situ breast cancer
* women with family high risk for breast cancer
* previous diagnosis of other cancers in the last 5 years
* early menopause women or in hormone replacement therapy

Ages: 44 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33200 (Estimated)
Dates: Start 2013-01; Primary Completion 2020-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of cumulative incidence of interval cancer cases by arm and by density group | three and six years
  An "interval cancer" is, according to European guidelines for quality assurance, a primary breast cancer which is diagnosed in a woman who had a screening test negative for malignancy within a time period equal to the screening interval. Interval cancers will be retrieved by linking the cancer registry and screening archive. The "cumulative incidence of interval cancers" is the number of interval cancers divided by the number of screened women
Comparison of cumulative incidence of T2+/node-positive status breast cancer cases by arm and by density group. | three and six years
  The "cumulative incidence of T2+/N+ breast cancer" is the number of cancers T2+/N+, regardless the modality of detection (screen-detected, interval cancer, etc.), divided by the number of screened women

SECONDARY OUTCOMES:
Comparison of false positive rates by arm and by density group | 3 and 6 years
  The "false positive rate" is measured as the sum of women with a positive mammography in a screening round without a breast cancer divided by the sum of screened women in the same round.
Comparison of cumulative incidence of breast cancer cases by arm and by density group. | 3 and 6 years
  The "cumulative incidence of breast cancer" is the cumulative number of breast cancers divided by the number of enrolled women.Breast cancer cases will be retrieved by linking the of enrolled women with cancer registry information
Comparison of attendance to mammography screening by arm and by density group. | 1, 2, 3, 4, 5 and 6 year
  The "attendance to mammography screening" is measured as the number of women attending screening mammography on the number of invited women.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Mantellini, MD, Principal Investigator — Cancer Prevention and Research Institute, ISPO
Locations (5):
- Italy (5):
  - Cancer Prevention and Research Institute, ISPO, Florence, FI
  - Local Health Unit, Forlì, Forlì-Cesena
  - CPO Piemonte, Torino, Torino
  - Local Health Unit n. 13, Mirano, Venezia
  - Local Health Unit n. 4, Thiene, Vicenza

REFERENCES:
- [Background] Kerlikowske K, Zhu W, Hubbard RA, Geller B, Dittus K, Braithwaite D, Wernli KJ, Miglioretti DL, O'Meara ES; Breast Cancer Surveillance Consortium. Outcomes of screening mammography by frequency, breast density, and postmenopausal hormone therapy. JAMA Intern Med. 2013 May 13;173(9):807-16. doi: 10.1001/jamainternmed.2013.307. PMID 23552817
- [Background] Paci E, Giorgi Rossi P. Tailored screening for breast cancer in premenopausal women: not just looking at sensitivity, but aiming to reduce burden. Womens Health (Lond). 2010 Jul;6(4):477-9. doi: 10.2217/whe.10.32. No abstract available. PMID 20597608
- [Background] Assi V, Warwick J, Cuzick J, Duffy SW. Clinical and epidemiological issues in mammographic density. Nat Rev Clin Oncol. 2011 Dec 6;9(1):33-40. doi: 10.1038/nrclinonc.2011.173. PMID 22143145
- [Background] Vachon CM, van Gils CH, Sellers TA, Ghosh K, Pruthi S, Brandt KR, Pankratz VS. Mammographic density, breast cancer risk and risk prediction. Breast Cancer Res. 2007;9(6):217. doi: 10.1186/bcr1829. PMID 18190724
- [Background] Pataky R, Ismail Z, Coldman AJ, Elwood M, Gelmon K, Hedden L, Hislop G, Kan L, McCoy B, Olivotto IA, Peacock S. Cost-effectiveness of annual versus biennial screening mammography for women with high mammographic breast density. J Med Screen. 2014 Dec;21(4):180-8. doi: 10.1177/0969141314549758. Epub 2014 Sep 3. PMID 25186116
- [Background] Blanch J, Sala M, Ibanez J, Domingo L, Fernandez B, Otegi A, Barata T, Zubizarreta R, Ferrer J, Castells X, Rue M, Salas D; INCA Study Group. Impact of risk factors on different interval cancer subtypes in a population-based breast cancer screening programme. PLoS One. 2014 Oct 21;9(10):e110207. doi: 10.1371/journal.pone.0110207. eCollection 2014. PMID 25333936
- [Background] Boyd NF, Huszti E, Melnichouk O, Martin LJ, Hislop G, Chiarelli A, Yaffe MJ, Minkin S. Mammographic features associated with interval breast cancers in screening programs. Breast Cancer Res. 2014 Aug 26;16(4):417. doi: 10.1186/s13058-014-0417-7. PMID 25346388
- [Background] Holm J, Humphreys K, Li J, Ploner A, Cheddad A, Eriksson M, Tornberg S, Hall P, Czene K. Risk factors and tumor characteristics of interval cancers by mammographic density. J Clin Oncol. 2015 Mar 20;33(9):1030-7. doi: 10.1200/JCO.2014.58.9986. Epub 2015 Feb 2. PMID 25646195
- [Background] Evans DG, Howell A. Can the breast screening appointment be used to provide risk assessment and prevention advice? Breast Cancer Res. 2015 Jul 9;17(1):84. doi: 10.1186/s13058-015-0595-y. PMID 26155950